CLINICAL TRIAL: NCT04934215
Title: Evaluation of Post-vaccination Anti-SARS-CoV-2 Serological Response in Health Care Workers With a History of COVID-19.
Acronym: VACCICOVID
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: VACCICOVID
Record Dates: First submitted 2021-06-17; First posted 2021-06-22 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: SARS CoV 2 Infection; Vaccination Reaction
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since the beginning of 2020, a major pandemic due to the new emerging coronavirus (SARS-CoV-2) has been spreading around the world. Today, the hope to contain this pandemic lies in the development and use of vaccines directed against this virus. Different strategies aim to maximize the early impact of vaccination in a context where few doses are available.

In early January 2021, large-scale vaccination began in France, first for populations at risk of severe COVID-19, but also for healthcare workers over 50 years of age or with an underlying pathology, and then for all voluntary healthcare workers.

DETAILED DESCRIPTION:
The question of vaccination of patients with a history of recent or late SARS-CoV-2 infection has rapidly become a major issue. Currently, French recommendations call for a single dose in the cohort that has been cured of COVID-19 for six months. In addition, the use of anti-SARS-Cov2 serology may be of interest because the presence of antibodies indicates recent or past contact with SARS-CoV-2. However, serological testing is not included in the vaccination decision strategy.

The goal of the investigators is to provide data on the immune response induced by SARS-CoV-2 vaccines in a real-world setting to support this choice. Given the absence of recommendations concerning the realization of the anti-SARS-CoV-2 serology, it will be proposed to all the nursing staff of the Groupe Hospitalier Paris Saint Joseph at the time of their vaccination, a serological screening.

The investigators will evaluate the dynamics of antibody production against the SARS-CoV-2 Spike protein after the first and second dose of vaccine (conventional prime-boost strategy recommended) in healthcare workers with or without a history of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Health care workers of the Paris Saint Joseph Hospital Group whose age ≥ 18 years
* French-speaking
* Health care workers who have received the BNT162b2 mRNA vaccine (COMIRNATY, Pfizer/BioNTech).

Exclusion Criteria:

* Health care workers under guardianship or curatorship
* Health care workers under court protection
* Health care workers who object to the use of their data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be carried out on the data of health care workers referred for vaccination to the Occupational Medicine Department and having received anti-SARS-CoV-2 serology at Day 21 post injection between 01/01/2021 and 31/03/2021, i.e. approximately 100 patients in total
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the level of serological response after the first and second vaccine doses in health care workers with and without a history of COVID-19. | Day 28
  Evolution of of anti-SARS-CoV-2 antibody level at D21-28 post-first dose and at D21-28 post-second dose in healthcare workers with and without a history of COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: PEAN DE PONFILLY Gauthier, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Marot S, Malet I, Leducq V, Zafilaza K, Sterlin D, Planas D, Gothland A, Jary A, Dorgham K, Bruel T; Sorbonne Universite SARS-CoV-2 Neutralizing Antibodies Study Group; Burrel S, Boutolleau D, Schwartz O, Gorochov G, Calvez V, Marcelin AG. Rapid decline of neutralizing antibodies against SARS-CoV-2 among infected healthcare workers. Nat Commun. 2021 Feb 8;12(1):844. doi: 10.1038/s41467-021-21111-9. PMID 33558507
- [Background] Dan JM, Mateus J, Kato Y, Hastie KM, Yu ED, Faliti CE, Grifoni A, Ramirez SI, Haupt S, Frazier A, Nakao C, Rayaprolu V, Rawlings SA, Peters B, Krammer F, Simon V, Saphire EO, Smith DM, Weiskopf D, Sette A, Crotty S. Immunological memory to SARS-CoV-2 assessed for up to 8 months after infection. Science. 2021 Feb 5;371(6529):eabf4063. doi: 10.1126/science.abf4063. Epub 2021 Jan 6. PMID 33408181
- [Result] Pean De Ponfilly G, Pilmis B, El Kaibi I, Castreau N, Laplanche S, Le Monnier A. Is the second dose of vaccination useful in previously SARS-CoV-2-infected healthcare workers? Infect Dis Now. 2021 Nov;51(8):673-675. doi: 10.1016/j.idnow.2021.07.001. Epub 2021 Jul 6. PMID 34242841